CLINICAL TRIAL: NCT07330349
Title: Influence of Alcohol, Psychoactive Drugs, and Analgesic Administration on the Evaluation Process in Patients With Penetrating Abdominal Trauma
Brief Title: Alcohol, Psychoactive Drugs, Analgesics and Evaluation in Penetrating Abdominal Trauma
Acronym: DIRECT
Status: Recruiting | Type: Observational
Sponsor: Fundacion Clinica Valle del Lili (Other)
Collaborators: Hospital Universitario del Valle Evaristo Garcia (Unknown)
Responsible Party: Principal Investigator, Alberto Federico García, Trauma and Acute Care Surgeon, Fundacion Clinica Valle del Lili
Other Study IDs: 2020.1639
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Injuries; Alcohol Intoxication; Substance-related Disorders; Penetrating Abdominal Trauma
Keywords: Trauma decision making; Time to surgery; Penetrating abdominal trauma; Alcohol use; Psychoactive substances; Analgesic administration
MeSH Terms: conditions — Abdominal Injuries; Alcoholic Intoxication; Substance-Related Disorders; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Penetrating Abdominal Trauma: Patients presenting with penetrating abdominal trauma who are evaluated and managed according to standard trauma care protocols, including immediate operative management or clinical observation with serial physical examination, as clinically indicated.
  Interventions: Other: Alcohol consumption; Other: Psychoactive substance use; Other: Analgesic administration

INTERVENTIONS:
Other: Alcohol consumption — Alcohol consumption prior to hospital admission, identified through patient report, clinical assessment, or laboratory testing when available, and observed as part of routine trauma care, not assigned by the study.
Other: Psychoactive substance use — Use of psychoactive substances prior to hospital admission, identified through clinical history, physical examination, or toxicology screening when available, and observed without modification by the study protocol.
Other: Analgesic administration — Administration of analgesic medications prior to or during initial hospital evaluation as part of standard trauma care, not assigned, standardized, or modified by the study.

SUMMARY:
This prospective observational study aims to evaluate whether alcohol consumption, psychoactive drug use, or prior administration of analgesics affects the clinical evaluation and surgical decision-making process in patients with penetrating abdominal trauma.

The study will be conducted in two level I trauma centers in Cali, Colombia: a public university hospital and a private university hospital, both with high volumes of trauma patients and established protocols for non-operative management using serial physical examination.

In many trauma centers, serial physical examination is used to safely identify patients who require surgical intervention. However, there is concern that intoxication or altered mental status may reduce the reliability of physical examination, potentially leading to unnecessary imaging studies, delays in surgical decision-making, or non-therapeutic laparotomies. Despite this concern, available evidence supporting these assumptions is limited.

Patients older than 14 years with penetrating abdominal trauma who undergo clinical evaluation to decide on surgical intervention. Patients will be classified according to the presence or absence of alcohol consumption, psychoactive substance use, or prior analgesic administration. The primary outcome is the time from hospital admission to the decision for surgical intervention. Secondary outcomes include trauma severity, need for surgery, length of hospital and intensive care unit stay, complications, and mortality.

By comparing patients with and without substance exposure across two different trauma care settings, this study seeks to determine whether serial physical examination remains a reliable and safe method for clinical decision-making in this population. The results may help optimize evaluation strategies, reduce unnecessary surgical procedures and diagnostic tests, and improve the standardization of care for patients with penetrating abdominal trauma.

DETAILED DESCRIPTION:
This is a prospective observational cohort study designed to evaluate the impact of alcohol consumption, psychoactive drug use, and prior administration of analgesics on the clinical evaluation process and surgical decision-making in patients with penetrating abdominal trauma.

The study will be conducted at two level I trauma centers in Cali, Colombia: one public university hospital and one private university hospital. Both institutions manage a high volume of trauma patients and apply standardized protocols based on serial physical examination for the evaluation of patients with penetrating abdominal trauma.

Patients older than 14 years who present with penetrating abdominal trauma and are hemodynamically stable will be evaluated according to routine institutional protocols, including serial abdominal physical examinations and selective use of diagnostic adjuncts such as focused abdominal sonography for trauma (FAST) or computed tomography, when clinically indicated. No additional diagnostic or therapeutic interventions will be performed as part of the study.

The exposure of interest is the presence of alcohol consumption, psychoactive substance use, or prior administration of analgesics before or during the initial clinical evaluation. These exposures will be identified through clinical assessment and medical record review and will be categorized according to predefined operational definitions.

The primary analytical focus is the interval between hospital admission and the decision for surgical intervention. Secondary analyses will explore associations between substance exposure and trauma severity, need for operative management, length of hospital stay, intensive care unit admission and length of stay, postoperative complications, and in-hospital mortality.

Data will be collected prospectively using standardized electronic case report forms. Data quality will be ensured through predefined range checks, consistency rules, and periodic review of entered data by the study investigators. Source data verification will be performed by comparing selected registry variables with information documented in the medical records.

Sample size was estimated to detect a clinically relevant difference in time to surgical decision between exposed and non-exposed patients, assuming an alpha level of 0.05, a statistical power of 80%, and an expected hazard ratio of 0.7. Based on the anticipated probability of requiring laparotomy of 0.68, a total of 247 events (laparotomies) were required, corresponding to 363 patients, to ensure an adequate number of events for time-to-event analysis.

Statistical analysis will include descriptive summaries of baseline characteristics, comparison of categorical variables using chi-square or Fisher's exact tests, and comparison of continuous variables using parametric or non-parametric methods as appropriate. Time-to-event analyses will be performed using Cox proportional hazards regression models, adjusting for relevant covariates such as age, sex, mechanism of injury, trauma severity, and type of substance exposure.

This study is observational and involves minimal risk to participants, as all evaluations and management decisions are part of standard clinical care. The results are expected to provide evidence regarding the reliability of serial physical examination in patients with penetrating abdominal trauma who present under the influence of alcohol, psychoactive substances, or analgesics, and may contribute to improving and standardizing trauma evaluation protocols across different clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency department with penetrating abdominal trauma.
* Age 14 years or older.
* Patients evaluated and managed according to standard trauma care protocols, including immediate operative management or clinical observation with serial physical examination, as clinically indicated.
* Patients admitted to the participating trauma centers during the study period.

Exclusion Criteria:

* Patients transferred from another institution after initial surgical intervention.
* Patients declared dead on arrival.
* Patients with incomplete or missing clinical data precluding assessment of outcomes of interest.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients aged 14 years and older presenting with penetrating abdominal trauma to two university-affiliated trauma centers in Cali, Colombia (one public and one private). Patients are evaluated and managed according to standard trauma care protocols, including immediate operative management or clinical observation with serial physical examination, as clinically indicated. The study assesses the impact of alcohol consumption, psychoactive substance use, and analgesic administration on the clinical evaluation process and surgical decision-making during hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 363 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Time to surgical decision | Up to 28 days
  Time elapsed from hospital admission to the clinical decision to proceed with surgical intervention, measured in hours, based on standard trauma care assessment.

SECONDARY OUTCOMES:
Need for surgical intervention | Up to 28 days
  Requirement of operative management during hospital stay.
Time to surgery | Up to 28 days
  Time elapsed from hospital admission to the start of surgical intervention, measured in hours.
In-hospital mortality | During hospitalization (Up to 28 days)
  Death occurring during the index hospitalization.
Trauma severity | 28 Days
  Trauma severity will be assessed using ATI (Abdominal trauma index).
Intraoperative bleeding | 28 days
  Intraoperative bleeding will be assessed by estimating total blood loss during the surgical procedure described by surgeon.

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Fundación Valle del Lili, Cali, Valle del Cauca Department
  - Hospital Universitario del Valle Evaristo García, Cali, Valle del Cauca Department

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Upon completion of the analysis and for up to five years thereafter
Access Criteria: Data will be shared on an individual basis with all individuals who make a reasonable request aimed at contributing to scientific knowledge